CLINICAL TRIAL: NCT05724225
Title: Atriogenic Tricuspid Regurgitation, Selected Omics Profile, Multimodality Imaging and Clinical Outcomes (the ATOMIC Study)
Brief Title: "Atriogenic Tricuspid Selected, Omics Profile, Multimodality Imaging and Clinical Outcomes"
Acronym: ATOMIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pedicino Daniela, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4424
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Tricuspid Valve Insufficiency
Keywords: functional tricuspid valve regurgitation; atrial fibrillation
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — samle blood to conduct an analysis and evaluate protein expression and Analysis of the correlation between circulating protein biomarkers and echocardiographic parameters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- First group with atrial fibrillation disease: 10 Atrial fibrillation(AF), predominant right atrial dilatation with at least moderate IT
- Second group with atrial fibrillation disease and tricuspid insufficiency: 10 AF, predominantly right atrial dilatation without TI (or TI no more than mild)
- Third group with AF and mitral insufficiency: 10 AF, predominantly left atrial dilatation with at least moderate MI
- Fourth group with atrial fibrillation and IM: 10 AF, predominantly left atrial dilatation without MI (or no more than mild MI)
- Fifth group with tricuspid insufficiency: 10 IT at least moderate to right ventricular remodeling in patients with pulmonary hypertension
- Sixth group with mitral insufficiency: 10 MI at least average from left ventricular remodeling from left ventricular dysfunction

SUMMARY:
The aim of our study is to investigate the molecular mechanisms underlying remodeling of the tricuspid valve apparatus in patients with ITF and isolated AF, in comparison with patients with ITF from right ventricular remodeling, patients with atriogenic MI and left ventricular remodeling. To achieve these aims, markers obtained from cardiovascular imaging methods, such as 3D echocardiogram, and biomarkers isolated from the peripheral blood of the study participants will be considered.

DETAILED DESCRIPTION:
Advances in echocardiography and, in particular, the development of three-dimensional echocardiography have allowed a more accurate analysis of the morphology of the tricuspid valve and a detailed understanding of the mechanisms underlying its insufficiency. From a clinical point of view, ITF is divided into a primary form, less frequent (8-10%), caused by primary alterations of the tricuspid valve apparatus, acquired or congenital, and in a "functional" form, the most frequent, conventionally associated in most cases with coexisting pathologies of the left heart or primitive pathologies of the right heart. More recently, long-lasting persistent atrial fibrillation (AF) has been associated with the development of ITF in the presence of structurally normal valve leaflets, preserved right ventricular size and function, and right atrial dilatation. This form of ITF, defined as "atrial functional", could benefit from a different therapeutic management compared to the classic form, more commonly caused by right ventricular dilatation and dysfunction ("ventricular functional" IT). However, not all patients with AF and tricuspid annulus dilatation develop valvular insufficiency and, on the other hand, with the same valvular annulus dilatation and right atrial size, the prevalence of severe IT forms is extremely variable.

This could depend on different adaptive mechanisms implemented by the valve leaflet tissue that lead to their growth or not in response to atrial remodeling and valve annulus dilatation, representing a key factor in the development and progression of the disease. Atriogenic ITF. If confirmed, these observations could lead to a better prognostic classification and different therapeutic perspectives for patients with AF at risk of developing forms of severe ITF and congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

- Admitted to the Department of cardiological, neurological and metabolic sciences of the San Luca hospital with a diagnosis of persistent atrial fibrillation

Exclusion Criteria:

* Patient aged <18 years;
* Pregnancy;
* Chronic inflammatory diseases;
* Autoimmune diseases;
* Tumor diseases;
* Chronic renal failure with eGFR < 30 mL/min;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with persistent atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Protein expression | 1 years
  Evaluation of the protein expression of the altered biomarkers in the 6 study groups

SECONDARY OUTCOMES:
Correlation between circulating protein biomarkers and diagnostic parameters | 6 months
  Analysis of the correlation between circulating protein biomarkers and echocardiographic parameters of mitral and tricuspid valve leaflet remodeling
Correlation between clinical data and diagnostic imaging markers | 6 months
  Evaluation of the correlation between clinical data (gender, age, AF duration) and echocardiographic imaging markers

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCSS Ospedale San Luca, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
All informtions about the patient is collected in a case report
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code